CLINICAL TRIAL: NCT03568669
Title: Neurocognitive Outcome as a Metric for Evaluating Therapeutic Intervention and Treatment Mechanisms in Congenital Central Hypoventilation Syndrome (CCHS): A Multi-Site Study Using The NIH Toolbox
Brief Title: Neurocognition in Congenital Central Hypoventilation Syndrome (CCHS)
Status: Recruiting | Type: Observational
Sponsor: Debra Weese-Mayer (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Seattle Children's Hospital (Other); Children's Hospital Los Angeles (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Debra Weese-Mayer, Professor of Pediatric Autonomic Medicine, Northwestern University Feinberg School of Medicine; Chief, Center for Autonomic Medicine in Pediatrics (CAMP), Ann & Robert H. Lurie Children's Hospital and Stanley Manne Children's Research Institute, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2016-167
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Congenital Central Hypoventilation Syndrome; Congenital Central Hypoventilation; CCHS; CCHS With Hirschsprung Disease; CCHS With Neural Crest Tumor; CCHS With Neuroblastoma
Keywords: NIH Toolbox; Toolbox; Congenital Central Hypoventilation Syndrome; CCHS; Autonomic Nervous System Dysregulation; PHOX2B
MeSH Terms: conditions — Congenital central hypoventilation syndrome; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NIH Toolbox Cognition Battery — An app-based cognitive assessment of executive function, attention, memory, and language that takes approximately 45 minutes to complete on an iPad

SUMMARY:
Congenital central hypoventilation syndrome (CCHS) is a rare disorder of autonomic and respiratory regulation that frequently alters oxygen delivery to the brain. In CCHS, neurocognitive function has been of great concern because of the potential for repeated hypoxemia and hypercarbia in activities of daily living in addition to hypoventilation with related hypoxemia and hypercarbia during sleep. As the world's leading referral center for CCHS, the Center for Autonomic Medicine in Pediatrics (CAMP) is engaged in ongoing research to identify factors that impact neurocognitive performance in patients with CCHS in order to optimize clinical management and improve long term neurocognitive outcomes.

The purpose of this IRB-approved research study is to implement the NIH Toolbox as a standard measurement of cognitive health in patients with CCHS. Further, the study aims to determine how intrinsic and extrinsic disease factors such as age at diagnosis, PHOX2B mutation type and genotype, and nature of past and present artificial respiratory intervention affect the NIH Toolbox Cognitive scores of individuals with CCHS. Eligible participants will complete a 45-minute NIH Toolbox assessment and parents (or adult participants) will complete an associated, 15-minute Research Electronic Data Capture (REDCap) questionnaire.

DETAILED DESCRIPTION:
CCHS is a genetic autonomic nervous system disorder caused by heterozygous mutations in the PHOX2B gene. 90-92% are caused by polyalanine repeat expansion mutations (PARMs) with 4 to 13 additional alanines on the affected allele in the 20 alanine repeat region of exon 3 (resulting genotype is 20/24-20/33). The remaining 8-10% of PHOX2B mutations are non-PARMs including missense, nonsense, frameshift or stop codon mutations. And less than 1% of CCHS patients are heterozygous for a large deletion eliminating the entire PHOX2B gene and potentially other neighboring genes. Different causative mutations vary in the level of associated protein dysfunction, leading to variability in the severity of the CCHS phenotype, and potentially in the severity and frequency of resulting neurocognitive insult. Severe cyanotic breath-holding spells and prolonged sinus pauses are two phenotypic features of CCHS known to alter regional blood flow/oxygen saturation to the brain (near-infrared spectroscopy; personal communication 2018). The fact that both of these phenotypic presentations are associated with particular PHOX2B genotypes suggests that genetic factors, intrinsic to CCHS pathology, might influence neurocognitive outcomes.

A recent report suggests that a number of extrinsic factors might also affect neurocognitive performance in patients with CCHS with later identification and less than conservative management in terms of artificial ventilation. While all cases of CCHS require assisted ventilation during sleep, some more severe cases require 24-hour/day artificial ventilation. Methods of assisted ventilation differ case-by-case and are chosen based on several factors, including the patient's level of alveolar hypoventilation, physician recommendation, and a family's ability to provide the recommended support. While these mechanisms are all meant to ensure optimal ventilation, the level of physiological oxygen stability and the stability of carbon dioxide levels provided with each varies. Thus, methods of respiratory assistance are likely to influence neurocognitive outcomes.

Currently, there is no standard mechanism for examining the neurocognitive impact that intrinsic pathology (PHOX2B genotype) and extrinsic factors (age of diagnosis and method of respiratory assistance) have on CCHS patients across age groups and between sites. In order to establish such a standard, this study aims to use a brief and reliable cognitive battery called the NIH Toolbox at multiple sites. The NIH Toolbox was developed to standardize evaluations in specific clinical populations for investigations of neurological development and change, disease recovery, and therapeutic interventions. The Toolbox consists of a series of cognitive assessments of executive function, attention, memory, and language designed for broad use across age groups from childhood to adulthood.

Participants in this study will initially be recruited during clinical visits at the Ann & Robert H. Lurie Children's Hospital of Chicago, Seattle Children's Hospital, and Children's Hospital Los Angeles as well as at meetings of the CCHS Family Network. All participants will complete a 45-minute NIH Toolbox cognitive assessment that is administered on an iPad by trained study staff. Additionally, parents (or adult participants) will complete a simple, 15-minute, electronic REDCap questionnaire designed to obtain basic information including PHOX2B genotype, age of CCHS diagnosis, past and present artificial ventilation interface (example mask, tracheostomy, etc.), past and present mode of artificial ventilation (positive pressure ventilator, negative pressure ventilator, phrenic nerve-diaphragm pacers), phenotype, and disease history. After initial participation, study subjects will complete the Toolbox and questionnaire at annual clinic visits or potentially at CCHS Family Network meetings to allow for longitudinal data collection.

The study will validate the NIH Toolbox as an assessment of cognitive performance and longitudinal cognitive outcomes in CCHS patients. Additionally, the study will characterize the effect of intrinsic and extrinsic disease factors on the neurocognitive outcomes of affected individuals in order optimize care for CCHS patients.

ELIGIBILITY:
Inclusion Criteria:

* PHOX2B mutation-confirmed CCHS diagnosis
* Speaks and reads English as a primary language

Exclusion Criteria:

* Unsuspected or unconfirmed CCHS
* Does not speak or read English as a primary language

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PHOX2B mutation-confirmed CCHS patients between 3-85 years of age, who speak and read English as a primary language.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Outcomes | January 2016 - December 2030
  Longitudinal neurocognitive outcomes in CCHS patients

SECONDARY OUTCOMES:
Neourcognitive Outcomes | January 2016 - December 2030
  Longitudinal neurocognitive outcomes based on participant age, PHOX2B genotype, and history of respiratory intervention

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington